CLINICAL TRIAL: NCT00732758
Title: Defining Vitamin D Insufficiency in School Age Children: A Randomized Placebo Controlled Trial of Vitamin D3
Acronym: Vitamin D RCT
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Kumaravel Rajakumar, Associate Professor of Pediatrics, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: 1K23HD052550-01A2 (NIH); 1K23HD052550-01A2 (NIH)
Record Dates: First submitted 2008-08-07; First posted 2008-08-12 (Estimated); Results first posted 2015-10-22 (Estimated); Last update posted 2015-12-29 (Estimated); Status verified 2015-11

CONDITIONS: Healthy
Keywords: Vitamin D Deficiency; Vitamin D Insufficiency; Child; Adolescent; African American; Caucasian; Definition; Preadolescent
MeSH Terms: conditions — Vitamin D Deficiency | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vitamin D3 (Experimental): Vitamin D3 1000 IU Tablet
  Interventions: Dietary Supplement: Vitamin D3 1000 IU
- Placebo (Placebo Comparator): Placebo Tablet
  Interventions: Dietary Supplement: Placebo Tablet

INTERVENTIONS:
Dietary Supplement: Vitamin D3 1000 IU — Vitamin D3 1000 IU Tablet once daily for 6 months
  Arms: Vitamin D3
Dietary Supplement: Placebo Tablet — Placebo Tablet once daily for 6 months
  Arms: Placebo

SUMMARY:
The study objective is to characterize the threshold levels of serum 25-hydroxyvitamin D for the definition of vitamin D insufficiency in 8-14 year old African American and Caucasian children.

We propose a 6 month randomized placebo controlled trial of vitamin D (vitamin D3 1000 IU/day vs. placebo) initiated during October through March (during fall and winter) in 8 to 14 year old African American and Caucasian children. The results of the trial will help establish the cutoff threshold value of serum 25(OH)D for defining vitamin D insufficiency in preadolescent and adolescent children. Safety of vitamin D supplementation will be assessed by measuring serum calcium at 0, 2 and 6 months and by monitoring for adverse events. Currently recommended adequate intake for vitamin D of 200 IU daily may not meet the body's daily needs for vitamin D. Therefore, it is likely that a higher level of daily vitamin D intake may be needed to meet the body's skeletal and non-skeletal demands for vitamin D. Determining the dietary required intake of vitamin D for the prevention of vitamin D insufficiency during childhood has immense public health potential for addressing health disparities and ensuring better bone health during adulthood. The primary outcome measure will be serum 25(OH)D and parathyroid hormone (PTH). The secondary outcome measures will include: markers of bone formation (serum P1NP) and bone resorption (serum CTX).We will also examine differences in serum 25(OH)D, PTH, and markers of bone turnover in African American vs. Caucasian children.

DETAILED DESCRIPTION:
Epidemiologic and clinical data document a high prevalence of vitamin D insufficiency among adults and adolescents in the US. Vitamin D insufficiency during childhood has the potential to impact the acquisition of peak bone mass. Vitamin D insufficiency is also associated with several non-skeletal disorders including cancer (prostate, breast, and colon), diabetes mellitus (type 1 and type 2), and multiple sclerosis. In our pilot study nearly 50% of 6 to 10 year old African American children residing in Pittsburgh, Pennsylvania, were deemed vitamin D insufficient (serum 25-hydroxyvitamin D (25(OH)D): ≤ 20 ng/mL; Rajakumar K, et al. Clinical Pediatrics. 2005;44:683-692). To extend this field further, we are proposing a randomized placebo-controlled trial of vitamin D3 for establishing the serum 25-hydroxyvitamin D (25(OH)D) cutoff threshold levels for defining vitamin D insufficiency during childhood and to document the safety and efficacy of treatment on the vitamin D status of the study cohort. A total of 168 (African American: 84, Caucasian: 84) 8 to 14 year old preadolescent and adolescent children will undergo a randomized-placebo controlled trial (RCT) of vitamin D3 1000 IU daily vs. placebo for 6 months initiated during fall and winter (October through March). Safety of vitamin D supplementation will be assessed by measuring serum calcium at 0, 2 and 6 months and by monitoring for adverse events. We will also examine the differences in serum 25(OH)D, PTH, and markers of bone turnover in African American vs. Caucasian children. The primary outcome measure will be serum 25(OH)D and PTH. The secondary outcome measures will include: markers of bone formation: serum osteocalcin (OC) and bone resorption: serum C-terminal cross-linking telopeptide of type 1 collagen (serum CTX). Additional outcomes will include: dietary intake of vitamin D and calcium, skin color (Fitzpatrick Sunreactive Skin Type and Melanin Index), sun exposure, and body mass index. Vitamin D deficiency will be defined as serum 25-hydroxyvitamin D concentrations <20 ng/mL. Public health importance of childhood vitamin D insufficiency is linked to the impact of vitamin D status on the acquisition of peak bone mass. Reduced peak bone mass can predispose to premature onset of osteoporosis and increase the risk for osteoporosis related fragility fractures. Achieving and maintaining vitamin D sufficiency during childhood can positively impact the skeletal health of children and reduce their "osteoporosis" burden during adulthood, and modify their risk for the non-skeletal disorders associated with chronic vitamin D insufficiency. Paucity of data regarding threshold levels of serum 25(OH)D associated with vitamin D insufficiency status among school age children and the likelihood that the serum 25(OH)D threshold levels for vitamin D sufficiency could be different among African American and Caucasian children makes it compelling for this issue to be explored. Based on expert opinion and supportive data in the medical literature, we feel that the currently recommended adequate intake for vitamin D for pre- and adolescent children (200 IU daily) is woefully inadequate to meet the daily needs for vitamin D. Therefore, it is likely that a higher level of daily vitamin D intake may be needed to meet the body's skeletal and non-skeletal demands for vitamin D. This study will determine the serum 25(OH)D cutoff for the definition of vitamin D insufficiency and document the safety and efficacy of treatment on vitamin D status.

ELIGIBILITY:
Inclusion Criteria:

* Age: 8-14 years
* Race: African American or Caucasian
* Children not taking multivitamins for at least 1 month before enrollment and agree not to start any multivitamin supplements during the 6-month trial period.
* Children who are on multivitamins can be considered for enrollment only if they are able to and agree to stop their multivitamin tablet for a 1 month washout period prior to enrollment.
* Absence of chronic diseases that could affect growth or calcium or vitamin D metabolism

Exclusion Criteria:

* Hepatic or renal disease
* Metabolic rickets
* Malabsorptive disorders (Crohn's disease, cystic fibrosis and celiac disease) or cancer
* Treatment with anticonvulsants or systemic glucocorticoids

Ages: 8 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 157 (Actual)
Dates: Start 2008-10; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kumaravel Rajakumar, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Result] Rajakumar K, Moore CG, Yabes J, Olabopo F, Haralam MA, Comer D, Bogusz J, Nucci A, Sereika S, Dunbar-Jacob J, Holick MF, Greenspan SL. Effect of Vitamin D3 Supplementation in Black and in White Children: A Randomized, Placebo-Controlled Trial. J Clin Endocrinol Metab. 2015 Aug;100(8):3183-92. doi: 10.1210/jc.2015-1643. Epub 2015 Jun 19. PMID 26091202

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We enrolled healthy 8- to 14-year-old children from October through March of 2008 through 2011.
Pre-assignment Details: Children receiving vitamin preparations underwent a 1-month washout before enrollment. Of 355 children assessed for eligibility, 304 were deemed eligible and among these 157 agreed to participate.
Groups:
- Vitamin D3 Group: Vitamin D3 1000 IU Tablet
  Vitamin D3 1000 IU: Vitamin D3 1000 IU Tablet once daily for 6 months
- Placebo Group: Placebo Tablet
  Placebo Tablet: Placebo Tablet once daily for 6 months
Period: Overall Study
Arm/Group | Vitamin D3 Group | Placebo Group
Started | 78 | 79
Completed | 70 | 63
Not Completed | 8 | 16
Not completed — Lost to Follow-up | 8 | 16

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vitamin D3 Group | Placebo Group | Total
Number analyzed (Participants) | 78 | 79 | 157
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.2 (1.9) | 11.4 (2.0) | 11.3 (1.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 34 | 79
  Male | 33 | 45 | 78
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 68 | 63 | 131
  Unknown or Not Reported | 9 | 15 | 24
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 42 | 42 | 84
  White | 36 | 37 | 73
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 78 | 79 | 157
Body Mass Index [Mean (Standard Deviation); unit: kilograms/meters^2] | 21.6 (5.5) | 21.6 (6.2) | 21.6 (5.85)
Skin Type [Number; unit: participants]
  I (easy burn, no tan) | 4 | 6 | 10
  II (easy burn, slight tan) | 14 | 13 | 27
  III (burn, then tan) | 15 | 16 | 31
  IV (no burn, good tan) | 36 | 27 | 63
  V (never burn, marked tan) | 7 | 16 | 23
  Unknown | 2 | 1 | 3
Vitamin D-deficient: Defined as serum 25(OH)D <20 ng/mL [Number; unit: participants]
  25(OH)D<20 ng/mL | 42 | 45 | 87
  25(OH)D>20 ng/mL | 36 | 34 | 70

OUTCOME MEASURES:

1. Primary Outcome: Serum 25-hydroxyvitamin D
Description: Circulating concentration of 25 hydroxyvitamin D is a biomarker of vitamin D status. Vitamin D deficiency was defined as serum 25-hydroxyvitamin D concentrations <20 ng/mL.
Time Frame: 6 months
Population: Intention to treat -- participants analyzed based on the group to which they were randomized but only included in the analysis if they had follow up data at 6 months.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Vitamin D3 Group | Placebo Group
Number analyzed (Participants) | 70 | 63
ng/mL | 26.7 (7.6) | 22.4 (7.3)
Statistical Analysis 1: Comparison: Vitamin D3 Group vs Placebo Group; Test type: Superiority or Other; p = 0.003, ANCOVA; adjusting for baseline 25(OH)D, race, BMI, diet vitamin D, gender, pubertal status, and sunlight exposure

2. Secondary Outcome: Parathyroid Hormone (PTH) Dietary Data
Time Frame: 6 months
Population: Intention to treat with participants analyzed by the group to which they were assigned but only analyzing those participants with follow up data for PTH at 6 months.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Vitamin D3 Group | Placebo Group
Number analyzed (Participants) | 69 | 62
pg/mL | 35.5 (16.3) | 33.5 (17.0)
Statistical Analysis 1: Comparison: Vitamin D3 Group vs Placebo Group; Test type: Superiority or Other; p = 0.51, t-test, 2 sided; unadjusted p-values

3. Secondary Outcome: Osteocalcin (OC)
Description: Marker of bone formation
Time Frame: 6 months
Population: Intention to treat with participants analyzed in the group to which they were assigned but only using participants with 6 month OC data available.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Vitamin D3 Group | Placebo Group
Number analyzed (Participants) | 70 | 61
ng/mL | 101.1 (48.3) | 104.8 (48.7)
Statistical Analysis 1: Comparison: Vitamin D3 Group vs Placebo Group; Test type: Superiority or Other; p = 0.66, t-test, 2 sided

4. Secondary Outcome: Collagen Type 1 Cross-linked C-telopeptide (CTx)
Description: Collagen type 1 cross-linked C-telopeptide (CTx) is a marker of bone resorption.
Time Frame: 6 months
Population: Intention to treat with participants analyzed by the group to which they were assigned but only analyzing participants with 6 month CTx data.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Vitamin D3 Group | Placebo Group
Number analyzed (Participants) | 69 | 63
ng/mL | 1.4 (0.9) | 1.6 (0.9)
Statistical Analysis 1: Comparison: Vitamin D3 Group vs Placebo Group; Test type: Superiority or Other; p = 0.35, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Vitamin D3 Group | Placebo Group
Serious Adverse Events (participants affected / at risk) | 0/78 | 0/79
Other Adverse Events (participants affected / at risk) | 0/78 | 0/79

LIMITATIONS AND CAVEATS:
No limitations.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No